CLINICAL TRIAL: NCT01769833
Title: HBsAg Decline and HBeAg Seroconversion Following 48 Weeks Peg-interferon-α Treatment in Patients With e Antigen Positive Chronic Hepatitis B After Nucleoside Analogue Maintenance Therapy Compared to Continuing Nucleoside Analogue Treatment
Brief Title: HBsAg Decline After Pegylated-interferon-α in e Antigen Positive Chronic Hepatitis B With Nucleoside Maintenance
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25659
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Hepatitis B
Keywords: HBsAg; Chronic hepatitis B; PEGinterferon Alfa-2A
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; Nucleosides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-interferon-alfa 2A (Active Comparator): PEG-interferon-alfa 2A
  Interventions: Drug: PEG-interferon-Alfa-2A
- Nucleosides (Placebo Comparator): Nucleosides
  Interventions: Drug: Nucleosides

INTERVENTIONS:
Drug: PEG-interferon-Alfa-2A — Pegasys ( PEG-interferon-Alfa-2A) 180mcg / subcutaneous / once-weekly
  Other Names: Pegasys (PEG-interferon-Alfa-2A)
  Arms: PEG-interferon-alfa 2A
Drug: Nucleosides
  Arms: Nucleosides

SUMMARY:
This study proposes to compare the effect of 48 weeks exposure to pegylated interferon alpha vs. nucleoside analogue (NA) on hepatitis B e antigen (HBeAg) seroconversion and HBsAg levels in nucleoside analogue controlled HBeAg-positive chronic hepatitis B (CHB) patients who have an undetectable hepatitis B virus (HBV) viral load at least 1 years.

DETAILED DESCRIPTION:
Pegylated interferon after long term NA therapy will potentiate the antiviral efficacy directly via its effect on broad antiviral activities and indirectly via activation of innate and adaptive immune responses leading to HBeAg seroconversion and eventually HBsAg loss and/or seroconversion.

This study proposes to compare the effect of 48 weeks exposure to pegylated interferon alpha vs. NA on HBeAg seroconversion and HBsAg levels in NA controlled HBeAg-positive CHB patients who have an undetectable HBV viral load at least 1 years.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age over 20 years
* HBeAg-positive CHB patients
* Patients treated with all available nucleoside analogue monotherapy or combination in Korea except telbivudine ( e.g.entecavir monotherapy or lamivudine/adefovir combination , lamivudine, adefovir monotherapy) for ≥ 18months and patients who have undetectable HBV viral load at least one year HBV DNA undetectable (≤ 400 copies/ml ) Serum alanine transferase: ≤ 10 X upper limit of normal (ULN) Baseline HBsAg: ≥ 102 IU/ml
* Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug. Additionally, all fertile males with partners of childbearing age and females must be using reliable contraception during the study and for 3 months after treatment completion.
* Obtaining written informed consent form

Exclusion Criteria:

* Decompensated cirrhosis or other contraindications to interferon alfa 2a therapy following local label.
* Concomitant or prior use of telbivudine.
* Positive test at screening for hepatitis A virus immunoglobulin M Ab, Hepatitis C virus-RNA or hepatitis C virus Ab, hepatitis delta virus Ab or HIV Ab.
* Diagnosed hepatic cellular carcinoma
* Any evidence of decompensated liver disease (Childs B-C)
* History or other evidence of a medical condition associated with chronic liver disease (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposures, thalassemia).
* Women with ongoing pregnancy or who are breast feeding.
* Evidence of alcohol and/or drug abuse within one year of entry.
* History of major organ transplantation with an existing functional graft.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
* Patients with a value of alpha-fetoprotein >100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months.
* patients having hypersensitivities for peginterferon alfa-2a or NAs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change in log10 HBsAg titer during antiviral therapy | 48 week
  To evaluate whether pegylated-IFNα2a treatment lowers HBsAg levels and eventually leads to HBsAg loss in patients after long term NA therapy compared to continuing NA treatment.

SECONDARY OUTCOMES:
HBV DNA undetectability and below 400 IU/mL during antiviral therapy and follow-up | 48 week, 96 week
HBeAg seroconversion and loss during antiviral therapy and at end of treatment and 1 and 2 years following end of treatment | 48 week, 96 week
HBsAg loss and HBsAg seroconversion at end of treatment and 1 and 2 years following end of treatment | 48 week, 96 week
Change in log10 HBsAg titer during follow-up | 48 week, 96 week
Mean change in log10 HBsAg titre over time, as estimated from the area between the baseline value and the curve of log10 HBsAg titre divided by the duration of treatment | 48 week

OTHER OUTCOMES:
effect of immune modulator therapy on the innate immune response in patients with HBeAg-positive CHB | 48 week, 96 week
  To evaluate the effect of immune modulator therapy on the innate immune response in patients with HBeAg-positive CHB in whom NA treatment has resulted in undetectable viral replication.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Heo, Dr, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

REFERENCES:
- [Derived] Woo HY, Heo J, Tak WY, Lee HJ, Chung WJ, Park JG, Park SY, Park YJ, Lee YR, Hwang JS, Kweon YO. Effect of switching from nucleos(t)ide maintenance therapy to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: A randomized trial. PLoS One. 2022 Jul 22;17(7):e0270716. doi: 10.1371/journal.pone.0270716. eCollection 2022. PMID 35867702